CLINICAL TRIAL: NCT02406482
Title: Evaluating a Microfinance Intervention for Vulnerable Women in Kazakhstan
Acronym: MFKZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Susan Witte, Associate Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAN8855; 5R01DA036514-03 (NIH)
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: HIV/AIDS and Infections
Keywords: sex work, Kazakhstan, microfinance, drug use
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections; Sex Work

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIVRR + MF (Experimental): Four sessions of education and intervention (Behavioral: HIV risk reduction (HIVRR)) followed by financial literacy, micro-savings and vocational training (Behavioral: Microfinance intervention (MF)).
  Interventions: Behavioral: Microfinance intervention (MF); Behavioral: HIV risk reduction (HIVRR)
- HIVRR only (Active Comparator): Four sessions of education and intervention (Behavioral: HIV risk reduction (HIVRR)).
  Interventions: Behavioral: HIV risk reduction (HIVRR)

INTERVENTIONS:
Behavioral: Microfinance intervention (MF) — Six sessions provided three times per week over two weeks by a study team facilitator. The sessions focus on banking services, savings (including how to open an account), budgeting (including development of a household budget), debt management, and financial negotiations, 1:1 matched savings account for women, followed by vocational training: Women assigned to the HIVRR+MF arm decide during their financial literacy sessions which vocational training program in which they would like to be enrolled (24 sessions).
  Arms: HIVRR + MF
Behavioral: HIV risk reduction (HIVRR) — Four sessions delivered twice a week for the first two weeks. Sessions derive from three evidence-based interventions with demonstrated efficacy to reduce drug and sexual HIV-risk behaviors in vulnerable women. Content focuses on basic transmission risk; educating about the risks of alcohol and drug use and how sexual behavior increases HIV risk; male and female condom use; examining the context for sexual risk including male partner sexual risk behavior (e.g. multiple partners) and violence against women; reducing other sexual risks (e.g., mutual masturbation, correct use of lubricants).

SUMMARY:
This study will examine the efficacy of a combined HIV and microfinance intervention to reduce biologically confirmed sexually transmitted infections (STIs), and new incidence of HIV and HCV, as well as reported sexual and drug risk behaviors among 520 women who have injected drugs in the past year and who engage in sex trading in Temirtau and Pavlodar, Kazakhstan. The proposed study builds on findings from an R34 by the investigative team testing a combination HIV prevention and microfinance intervention. Building on successful protocols and significant results, we will randomly assign 520 women who inject drugs and engage in sex trading from Temirtau and Pavlodar, Kazakhstan to either (1) a 4 session HIV prevention intervention combined with a 6 session financial literacy intervention, enrollment in an existing vocational training program and receipt of matched savings (HIVRR+MF); or to the 4 session HIV prevention intervention alone. The HIVRR intervention is guided by social cognitive theory. The HIVRR+MF intervention integrates asset theory with social cognitive theory. The MF includes: 1) financial literacy; 2) vocational training; and 3) micro-savings to support transition to a more permanent employment status. We hypothesize that increasing financial literacy, enhancing vocational skills required to fill marketable positions in the local economy, and beginning a personal savings program, combined with HIV risk reduction, will lead to significant reductions in study outcomes compared to an HIVRR intervention without a microfinance intervention.

DETAILED DESCRIPTION:
1. STUDY PURPOSE AND RATIONALE. This study is a 2-arm randomized control clinical trial (RCT), Project Ascension, that will evaluate the efficacy of a combined 4-session HIV risk reduction and microfinance intervention (including 6 sessions of financial literacy skills; referral to a 36 session vocational training; and concurrent weekly matched savings from the research team) (HIVRR+MF) to reduce new HIV/STI infections and sexual and drug risk among women who inject drugs and trade sex in Temirtau and Pavlodar, Kazakhstan. The primary outcomes are to decrease new STIs, including HIV and HCV, proportion of unprotected sexual acts and proportion of income from sex work. Secondary outcomes include examining mediating and moderating factors, the examine women's experience of the intervention and cost effectiveness of the addition of MF over HIVRR alone on primary outcomes.

   To evaluate the impact of the HIVRR+MF intervention we will use two sources of data: (1) individual level biological testing data for syphilis, gonorrhea, trichomonas, HIV and HCV collected from 520 participants, randomly assigned to either the treatment arm or control arm at baseline, 6-months post-intervention, and 12 months post-intervention; and (2) self-reported data collected from participants at baseline, 3 months-, 6 months-, and 12 months post-intervention. The same outcomes and variables will be collected at each time point.

   We are also currently seeking approval for this study from the IRB at the Kazakh School of Public Health.
2. STUDY DESIGN AND STATISTICAL PROCEDURES.

This RCT will be conducted with 520 FSW-PWID recruited from 2 NGOs, one each in Temirtau and Pavlodar, Kazakhstan. Collaborating NGOs are You are Not Alone, in Pavlodar and the Association of People Living with HIV in Temirtau. They provide the full spectrum of services for people affected by STIs and HIV, including FSW-PWID in each city. Women will be randomly assigned to either a (1) HIVRR plus Microfinance (HIVRR+MF) or (2) HIVRR alone control condition. We will compare two active conditions offering the HIV risk reduction intervention (HIVRR) to both intervention arms. This design will allow us to examine how the addition of the MF to HIVRR might lead to superior outcomes compared to receiving HIVRR alone. HIVRR intervention and the financial literacy will be delivered by research staff and vocational training will be delivered by field site staff. In month 6, recruitment will begin. We will enroll an average of 22 women per cohort per site (44 total every 2.5 months) and complete enrollment by month 35. Self-reported data on behavioral outcomes will be collected via audio computer-assisted self-interview (ACASI) and assessed at baseline, 3, 6, and 12 months post-intervention. We will implement the same survey at each time point. Primary outcomes will be measured via biological assay for Neisseria gonorrhea, Trichomoniasis, Syphilis, Chlamydia and Mycoplasma, as well as for HIV and HCV. Biological outcomes are assessed at baseline, 6 and 12 months post-intervention. Follow up assessments will start in month 15 and the final 12 month follow up will be completed in month 51. For Aim 4, we will conduct a qualitative study on women's experience with each of the HIVRR+MF components, and the unique impact of study conditions on structural factors associated with risk among FSW-PWID. For Aim 5, we will collect cost data related to each intervention component every 6 months from months 6-50. Data analyses will commence in year 5 followed by dissemination of findings.

Qualitative Study. To help open the "black box" of the delivery of HIVRR+ MF, the investigators will conduct semi structured in-depth interviews at 3 points in time during implementation of the HIVRR intervention. Following the HIVRR and financial literacy components (4 weeks post-baseline), investigators will randomly select 2 participants from each arm per cohort (total of N=48 women from 12 cohorts) to complete their first of 3 interviews. The next two interviews will be conducted at the end of the MF intervention and again at the 12 month follow up for each participant. Questions will focus on participants' perception of the intervention, their experience receiving the intervention components (including reactions or interactions with family, friends, colleagues related to their participation), their experience receiving the sessions, factors promoting the use of the session information and skills and barriers impeding participation. Importantly, questions will also focus on perceptions of how the intervention influenced participant safety, including any policy involvement, stigma or discrimination, drug use before and during the intervention, and savings and the potential access to matched savings. All interviews will be audio taped, transcribed and translated to English.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years old;
2. reports having engaged in vaginal or anal sexual intercourse in the past 90 days in exchange for money, alcohol, drugs, or other goods;
3. reports having injected drugs in the past year;
4. reports having engaged in unprotected sexual intercourse in the past 90 days with either a paying, casual, or intimate (main) sexual partner;
5. reports being interested in learning a marketable vocation, specifically hairdressing or cooking/baking.

Exclusion Criteria:

1. assessed to have a severe cognitive or psychiatric impairment that would interfere with the ability to provide informed consent or complete study instruments. (As in prior SIG and GHRCCA studies, a standardized diagnostic tool will not be used. Rather, as part of informed consent, a potential participant is asked to state her understanding regarding three areas covered earlier during the informed consent protocol: (a) the nature and extent of participation in the study; (b) the risks involved with participation; and (c) the potential benefits of participation in the study. If a participant is unable to respond to any of the three items by reiterating the information presented earlier, she will be excluded from the study.)
2. does not speak and understand Russian at a conversational level;
3. unwilling or unable to commit to completing the study;
4. has plans to move two or more hours away from the study site during the study follow up period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2015-04; Primary Completion 2018-08-01 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Incidence of biologically confirmed STIs | 12 months
  To examine whether women assigned to the combined HIVRR+MF intervention have: (1) a lower cumulative incidence of biologically confirmed STIs syphilis, gonorrhea, chlamydia trichomoniasis and mycoplasma)
Rate of new HIV and HCV cases | 12 months
  To examine if the rate of new HIV and HCV cases is lower compared to those assigned to the HIVRR arm over the 12 month follow-up
Number of unprotected vaginal and anal sexual acts with both regular and paying partners | 12 months
Proportion of unprotected vaginal and anal sexual acts with both regular and paying partners | 12 months
Number of unsafe injection acts | 12 months
Proportion of unsafe injection acts | 12 months
Proportion of monthly income from sex work | 12 months
  To examine whether there is a lower proportion of monthly income from sex work at 3, 6, and 12 months, compared to women assigned to HIVRR

CONTACTS AND LOCATIONS:
Overall Officials: Susan Witte, Ph.D., Principal Investigator — Columbia University
Locations (3):
- Kazakhstan (3):
  - GHRCCA office, Almaty
  - GHRCCA office, Pavlodar
  - GHRCCA office, Temirtau

REFERENCES:
- [Derived] Mukherjee TI, Terlikbayeva A, McCrimmon T, Primbetova S, Mergenova G, Benjamin S, Witte S, El-Bassel N. Association of gender-based violence with sexual and drug-related HIV risk among female sex workers who use drugs in Kazakhstan. Int J STD AIDS. 2023 Sep;34(10):666-676. doi: 10.1177/09564624231170902. Epub 2023 Apr 21. PMID 37083464
- [Derived] El-Bassel N, McCrimmon T, Mergenova G, Chang M, Terlikbayeva A, Primbetova S, Kuskulov A, Baiserkin B, Denebayeva A, Kurmetova K, Witte SS. A cluster-randomized controlled trial of a combination HIV risk reduction and microfinance intervention for female sex workers who use drugs in Kazakhstan. J Int AIDS Soc. 2021 May;24(5):e25682. doi: 10.1002/jia2.25682. PMID 33955170
- [Derived] McCrimmon T, Witte S, Mergenova G, Terlikbayeva A, Primbetova S, Kuskulov A, Bellamy SL, El-Bassel N. Microfinance for women at high risk for HIV in Kazakhstan: study protocol for a cluster-randomized controlled trial. Trials. 2018 Mar 20;19(1):187. doi: 10.1186/s13063-018-2566-y. PMID 29558982